CLINICAL TRIAL: NCT05141136
Title: A Magnetic Resonance Imaging Study of the Spread of Local Anesthetic Solution in Patients Receiving Ultrasound-guided Paravertebral Block at the Thoracic 2 Spinal Level: Prospective Randomized Controlled Study
Brief Title: Magnetic Resonance Imaging of Injectate in Thoracic 2 Paravertebral Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3-2021-0293
Record Dates: First submitted 2021-09-27; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Cervical Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: Patients with chronic cervical radiculopathy due to degenerative spinal disease for more than 3 months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Medical staff performing patient care, including pain management, and investigators who investigate and record observations and evaluations, and those who analyze magnetic resonance imaging, are kept unaware of group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound probe sagittal group (Experimental): A thoracic 2 paravertebra block is performed with the ultrasound probe placed sagittal and the needle in plane with respect to the probe.
  Interventions: Procedure: Ultrasound probe sagittal group
- Ultrasound probe transverse group (Active Comparator): A thoracic 2 paravertebra block is performed with the ultrasound probe placed transverse and the needle in plane with respect to the probe.
  Interventions: Procedure: Ultrasound probe transverse group

INTERVENTIONS:
Procedure: Ultrasound probe sagittal group — Place the ultrasound probe vertically against the patient's spine and insert the needle in-plane. The width of insertion of the needle is usually approximately 5 cm from the midline. After the needle penetrates the superior costovertebral ligament and pops, when it reaches the thoracic paravertebral space, perform aspiration and inject 10 mL of 1% lidocaine. At this time, it can be observed in real time as the infusion fluid pushes the bright pleura away from the needle.
  Arms: Ultrasound probe sagittal group
Procedure: Ultrasound probe transverse group — Place the ultrasound probe transverse to the spine and insert the needle in-plane. The reflection of a transverse process is a common landmark. The needle goes in from lateral to in plane. The goal is a triangle between the parietal pleura anteriorly and the internal intercostal membrane and intercostal muscle posteriorly. The final point of the needle is the transition zone from the intercostal to the thoracic paraspinal space, just anterior to the transverse process. When it is confirmed that the tip of the needle has reached the paravertebral space, 10 mL of 1% lidocaine is injected after checking the negative pressure, and after confirming the spread of the drug in real time with ultrasound.
  Arms: Ultrasound probe transverse group

SUMMARY:
The purpose of this study is to analyze the spread of local anesthetic using magnetic resonance imaging after thoracic 2 paravertebral block in patients with cervical radiculopathy.

DETAILED DESCRIPTION:
1. Ultrasound guided thoracic 2 paravertebral block will be done using sagittal scan or transverse scan.
2. Clinical parameters will be monitored (temperature, perfusion index, assessment of sensory block and analgesic effect, vital sign, adverse events) after the nerve block.
3. Cervical MRI will be taken 1 hour after the nerve block.
4. Follow up 7 days and 28 days after the MRI at outpatient clinic (numeric rating scale, medication quantification scale)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral radiating pain in the upper extremity whose pain persists for more than 3 months despite conservative treatment
2. Diagnosis: cervical degenerative disc disease, cervical foraminal stenosis, cervical stenosis with/without myelopathy
3. Numeric rating score ≥ 4
4. 19 years or older

Exclusion Criteria:

1. Cervical or upper thoracic spine surgical history
2. If the body mass index is 35 kg/m2 or more
3. If you have an allergy or hypersensitivity reaction to a local anesthetic
4. coagulation disorders
5. Local infection at the injection site
6. claustrophobia
7. If you have a metal insert such as a pacemaker
8. pregnancy
9. Patients who are unable to communicate and have cognitive impairment
10. If a person who cannot read the consent form is included among the subjects (e.g., illiterate, foreigners, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Injectate spread on MRI imge | 1 hour after thoracic 2 paravertebral block
  Presence of injectate on each anatomic target (Paravertebral space, ventral/dorsal epidural space, intercostal nerve, contralateral space)

SECONDARY OUTCOMES:
numeric rating score | Before nerve block, after 30 minutes, and thereafter, at the outpatient visit on the 7th day and the outpatient visit on the 28th day.
  A score of 0 indicates no pain and a score of 10 indicates maximum pain.
perfusion index | Before nerve block, after 30 minutes
  After the subject rests in the supine position for about 10 minutes, pulse oximetry is placed on the index finger to record the baseline value. Perfusion index was measured using pulse oximetry (Root®, Masimo Corporation, Irvine, CA, USA). The perfusion index can be a useful indicator for judging the After the subject rests in the supine position for about 10 minutes, pulse oximetry is placed on the index finger to record the baseline value. Perfusion index was measured using pulse oximetry (Root®, Masimo Corporation, Irvine, CA, )
skin temperature | Before nerve block, after 30 minutes
  Place a touch thermometer (IntelliVue MP70 patient monitor, Philips Healthcare, Best, Netherlands) on the palm of your hand and measure. Calculate the amount of change from the baseline. Record the difference with the contralateral hand.
pinprick and cold test | Before nerve block, after 30 minutes
  Pinprick sensation was performed using a 22 gauge short bevel needle. Comparison with the contralateral dermatome. Sensation is rated as 0 (no sensation), 1 (decreased sensation), and 2 (normal). A sensory block is considered successful if the patient reports 0 or 1. Cold sensation is measured in the same way using an ice cube. If there is no difference in the sensation of the treated dermatome compared to the contralateral dermatome.
Blood pressure in mmHg | Before nerve block, after 30 minutes
  Record blood pressure , and calculate the change from baseline.
Pulse rate in /min | Before nerve block, after 30 minutes
  Record pulse, and calculate the change from baseline.
Presence of adverse events | Before nerve block, after 30 minutes
  Horner syndrome, hoarseness, dyspnea, ptosis, dysphagia
medication quantification scale | Before nerve block, and thereafter, at the outpatient visit on the 7th day and the outpatient visit on the 28th day
  The Medication Quantification Scale (MQS) is an instrument with potential clinical and research applications for quantifying medication regimen use in chronic pain populations.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No